CLINICAL TRIAL: NCT02139722
Title: A Patient-Centered Intervention to Increase Screening of Hepatitis B and C Among Asian Americans
Brief Title: Patient-Centered Care and Asian Americans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: San Francisco Hep B Free Campaign (Unknown); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: AD-11-4615
Record Dates: First submitted 2014-05-06; First posted 2014-05-15 (Estimated); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Hepatitis B; Hepatitis C; Liver Disease
Keywords: hepatitis B; hepatitis C; screening; Asian Americans; mobile technology
MeSH Terms: conditions — Hepatitis B; Hepatitis C; Liver Diseases

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Provider Panel Notification (PPN) Alone (No Intervention): The comparison procedures consist of a panel notification given to providers and an audio-visual presentation on diet and exercise given to patients.
- Video Doctor, PA + PPN (Experimental): Video Doctor (VD) and Provider Alert (PA) intervention combined with Provider Panel Notification (PPN)
  Interventions: Behavioral: Video Doctor, PA + PPN

INTERVENTIONS:
Behavioral: Video Doctor, PA + PPN — The intervention consists of a Video Doctor and Provider Alert. For the Video Doctor, we will develop a series of 30-60 seconds video clips, a branching algorithm, and a mobile application linking the baseline survey to the clips. The Provider Alert is a point-of-care reminder printout generated by the mobile application to facilitate patient-provider communication. The intervention integrates guidelines, literature, guidance from the Systems Model, our prior work, and input from patients and providers.
  Arms: Video Doctor, PA + PPN

SUMMARY:
Liver cancer and hepatitis B are health disparities for Asian Americans, and hepatitis C is a rising problem. Little is known about how to improve the quality of health care Asian Americans receive for viral hepatitis. Technology, specifically mobile applications, can provide a flexible and efficient way to address these challenges. This project seeks to develop, implement, and test an intervention to increase hepatitis B and C screening for Asian Americans in 2 healthcare systems in San Francisco.

The research team will develop, implement, and evaluate the efficacy of an interactive, patient- centered mobile app for use on a tablet computer to increase hepatitis B and C screening among unscreened Asian Americans age 18 and older. The team will use their experience in health promotion to develop the intervention by working with patients, community leaders and advocates, clinical staff, healthcare providers, and healthcare system administrators from a county safety net system and an academic primary care practice in the San Francisco Bay Area. The mobile application will include video clips with a physician (Video Doctor) addressing patient concerns regarding hepatitis B and C screening in the patient's preferred language, English, Chinese, or Vietnamese. A patient who has not been screened for hepatitis B will answer questions about his or her characteristics and preferences using the mobile application. The mobile application will then show 30-60 seconds video clips with messages that address the patient's responses related to hepatitis B screening and that are delivered by an actor playing a physician. Those who are born between 1945 and 1965 also receive messages about hepatitis C screening. At the end, the tablet computer will generate a provider alert to let the treating provider know what the patient's preferences are regarding testing for viral hepatitis.

Once developed, the intervention will then be used in combination with a physician panel notification and tested against physician panel notification only in a randomized controlled trial to see which approach is better in increasing the rate of hepatitis B and C screening. The team will also work with the 2 healthcare system to ensure that the interventions will be practical and easily adopted once the study is over. The findings of this project will greatly expand understanding about how to use technology- based interventions to improve quality of healthcare in diverse patient populations.

ELIGIBILITY:
Inclusion Criteria:

* ages 18+ years
* identifies as Asian
* Asian American, Chinese, or Vietnamese
* speaks English, Chinese (Cantonese), or Vietnamese
* does not have an electronic health record (EHR)-documented HBV screening test (defined as a hepatitis B surface antigen [HBsAg] test).
* we select Chinese and Vietnamese because those are the 2 most common languages spoken by limited English-proficient Asian Americans

Exclusion Criteria:

* dementia or any conditions precluding understanding informed consent or using a touch screen with audio

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 431 (Actual)
Dates: Start 2014-01-02 (Actual); Primary Completion 2017-05-28 (Actual); Study Completion 2017-07-30 (Actual)

PRIMARY OUTCOMES:
EHR-documented hepatitis B surface antigen (HBsAg) test | 3 months
  The main outcome measure is an EHR-documented hepatitis B surface antigen (HBsAg) test at 3 months post-intervention. We chose screening for hepatitis B because, among adults, particularly immigrants or descendants of immigrants, it is the most important first step in the control of viral hepatitis B and lack of screening remains a significant problem. While many young adult Asian Americans born in the U.S. or who immigrated at a young age may have been vaccinated for hepatitis B as a child or prior to entering college, pre-vaccination testing may not have been done. Given the high rates of infection in their parents and the possibility of vertical transmission, all Asian Americans should be tested for chronic hepatitis B using the HBsAg test. All screening outcomes (test receipt) as well as test ordering by the healthcare providers will be collected from the medical record through the EHRs at 3-month post-intervention.

SECONDARY OUTCOMES:
Knowledge about hepatitis B virus (HBV) and hepatitis C virus (HCV) | 3 months
  Data sources include the self-administered pre-intervention survey via a tablet computer, and the post-intervention phone survey administered by a research assistant, and EHR. All patient surveys will be done in the patient's preferred language (English, Chinese, or Vietnamese). Pre- and post-intervention survey data of secondary outcomes include: Knowledge (awareness of HBV and HCV, screening test, modes of transmission); Self-efficacy (perceived confidence in initiating conversation and request screening test from providers); Patient-Provider Communication Experiences (asked provider for HBV or HCV test, discussed HBV or HCV test with provider, receipt of provider recommendation to get a HBV or HCV test).

CONTACTS AND LOCATIONS:
Overall Officials: Tung T Nguyen, MD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - Zuckerberg San Francisco General, San Francisco, California
  - University of California, San Francisco, San Francisco, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Khalili M, Kim NJ, Tsoh JY, Walsh JME, Goldman LE, Gildengorin G, Wong C, Tran MT, Yu E, Sharp MT, LeTran VH, Nguyen VV, Nguyen TT. Health Within Reach-a Patient-Centered Intervention to Increase Hepatitis B Screening Among Asian Americans: a Randomized Clinical Trial. J Gen Intern Med. 2022 Oct;37(13):3242-3250. doi: 10.1007/s11606-021-07232-3. Epub 2022 Jan 6. PMID 34993863